CLINICAL TRIAL: NCT04307433
Title: mHealth Delivered Narrative Intervention to Increase Cervical Cancer Screening Among Malawian Women Living With HIV
Brief Title: Storytelling Intervention to Promote Cervical Cancer Screening Uptakes Among Malawian Women Living With Human Immunodeficiency Virus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Boston (Other)
Responsible Party: Principal Investigator, Haeok Lee, Professor, University of Massachusetts, Boston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019250
Record Dates: First submitted 2020-03-10; First posted 2020-03-13 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: The proposed study has two phases:
  Phase 1. Development of Narrative Video: The investigators will first develop culturally-grounded and human-centered storytelling narrative intervention videos in Chichewa, the local language to address sociocultural and individual factors which influence cervical cancer prevention behaviors. The video will be filmed in person in community organizations in Malawi.
  Phase 2: A Pilot Randomized Controlled Trial (RCT) of a Story Telling Narrative Intervention: The investigators will conduct a three-arm pilot RCT using the storytelling-based intervention delivered by mHealth (tablets) with 180 women residing in a rural community in Malawi. The intervention groups (Arm 1: storytelling narrative video on tablets [n=60] & Arm 2: a video with a voice over presenting didactic materials on tablets [n=60]) will watch approximately 30 minutes of video intervention and the comparison group (Arm 3 [n=60]) will be read non-narrative educational materials
Who Masked: Outcomes Assessor
Masking Description: The data collector who assesses the follow-up assessments will be blind to treatment condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): ST Narrative + mHealth: Storytelling narrative video on tablets
  Interventions: Behavioral: Storytelling narrative videos on tablets
- Arm 2 (Active Comparator): mHealth: a video with a voice over presenting didactic materials on tablets
  Interventions: Behavioral: Storytelling narrative videos on tablets
- Arm 3 (Placebo Comparator): Control: non-narrative educational materials will be read
  Interventions: Behavioral: Storytelling narrative videos on tablets

INTERVENTIONS:
Behavioral: Storytelling narrative videos on tablets — The storytelling narrative episodes in the application will feature video clips of the multiple stories of women living with HIV infection, HIV support group leaders, community leaders, and health care professionals and a Learn More video of physician discussing cervical cancer.

SUMMARY:
To develop a theory-based culturally-grounded storytelling-based intervention to increase cervical cancer screening among Malawian women living with HIV infection. Secondary objectives: To conduct a pilot randomized clinical trial (RCT) to examine the acceptability, feasibility and preliminary effectiveness of narrative intervention on cervical cancer screening prevention behavior.

DETAILED DESCRIPTION:
Design

This two year project will employ a holistic community-based approach for recruitment. The project will involve two phases: Phase 1: The investigators will produce culturally-grounded and human-centered storytelling narrative intervention videos to address sociocultural and individual factors which influence cervical cancer prevention behaviors. Phase 2: The investigator will conduct a pilot RCT using the storytelling-based intervention delivered by mHealth (tablets) with 180 women residing in a rural community in Malawi. The intervention groups (Arm 1: storytelling narrative video on tablets [n=60] & Arm 2: a video with a voice over presenting didactic materials on tablets [n=60]) will watch approximately 30 minutes of video intervention and the comparison group (Arm 3 [n=60]) will be read non-narrative educational materials. Study measures of attitudes, knowledge, and cervical cancer screening intention will be assessed by pre-test and immediate post-test interviews, then again at 2 and 6-months following the intervention.

Selection and Enrollment

Inclusion criteria are: 1) being confirmed HIV positive based on medical records, 2) women living with HIV infection (WLHIV) support group members, 3) ages 20-50 years, 4) no prior cervical cancer screening, 5) no history of invasive cervical cancer, and 6) willingness to participate in the study. The age range to 20-50 years for cervical cancer screening because there is limited evidence that this is the optimal upper age for cervical cancer screening of HIV-infected women (World Health Organization [WHO] 2013).

This study will use a sequential-stratified sampling method. Of the eligible support groups and among those expressing interest, the investigators will select 15 support groups from rural areas within the Lilongwe district and then randomly assign the selected groups into intervention and comparison arms. The computer-generated assignments will be stratified by support group size and the distance between intervention and control arms (at least 4 miles). Within each selected support group, 12 women who are eligible will be invited to participate in the study. The investigators have satisfactorily used these methods for recruitment of WLHIV by working with HIV support group leaders in our previous studies.

ELIGIBILITY:
Inclusion Criteria:

Women who:

1. are confirmed HIV positive based on medical records
2. are women living with HIV infection support group members
3. are ages 20-50 years
4. are no prior cervical cancer screening
5. are no history of invasive cervical cancer
6. are willingness to participate in the study

Exclusion Criteria:

1. are not able to speak Chichewa or English
2. self-report currently receiving treatment of a serious mental illness (e.g., schizophrenia and bipolar disorder)

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — females are biologically eligible because the research involves cervical cancer prevention. Inclusion of males in the study would be inappropriate due to lack of cervical cancer incidence.
Enrollment: 179 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Number of Participant with Cervical Cancer Screening Uptakes | six months post-intervention
  will be measured through self-report and health passport record review

CONTACTS AND LOCATIONS:
Overall Officials: Haeok Lee, PhD, Principal Investigator — University of Massachusetts, Boston
Locations (1):
- Community organization, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: No